CLINICAL TRIAL: NCT01966549
Title: A Randomized, Placebo Controlled Double-Blind, Multi-Center, Phase II Study to Assess the Efficacy and Safety of CNTO6785 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Effectiveness and Safety of CNTO6785 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102318; CNTO6785OPD2001 (Other: Janssen Research & Development, LLC); 2012-003607-36 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Moderate to Severe Chronic Obstructive Pulmonary Disease; CNTO 6785; Placebo
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNTO 6785 (Experimental)
  Interventions: Drug: CNTO 6785
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTO 6785 — CNTO 6785 (6 mg/kg) will be administered by intravenous (into a vein) infusion on Weeks 0, 2, 4, 8 and 12. Participants who weigh more than 100 kg will receive a dose of 600 mg of CNTO 6785.
  Arms: CNTO 6785
Drug: Placebo — Sterile, 5 percent dextrose will be used as the placebo in this study. Placebo will be administered by intravenous infusion on Weeks 0, 2, 4, 8 and 12.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of CNTO6785 compared with placebo in participants with moderate to severe Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
This is a multi-center, randomized (study medication is assigned by chance), placebo-controlled (effect of the study medication will be compared with the effect of placebo [inactive substance]), double-blind (neither physician nor participant knows the treatment that the participant receives), parallel-group study (each group of participants will be treated at the same time). This study consists of 3 phases: a screening phase (within 3 weeks prior to the start of study medication), a treatment phase (12 weeks), and a follow-up phase (12 weeks after the last administration of study medication). Approximately 170 participants will be enrolled in this study to receive CNTO6785 or placebo in 1:1 ratio. Safety will be evaluated by the assessment of adverse events, vital signs, 12-lead electrocardiogram, physical examination, early detection of active tuberculosis, and clinical laboratory tests which will be monitored throughout the study. The total duration of study participation for a participant will be 30 weeks.

ELIGIBILITY:
Inclusion criteria:

* Moderate to severe Chronic Obstructive Pulmonary Disease (COPD) (Grade II or Grade III according to the GOLD Guidelines) with chronic bronchitis (sputum production on most days for at least 12 weeks per year for at least 2 successive years) at screening
* Persistent COPD symptoms that required repeated (greater than 1) 'as needed' use of a short acting rescue medication within 4 weeks prior to screening
* Had at least 2 COPD exacerbations requiring antibiotics and/or systemic corticosteroids in the past 2 years OR able to spontaneously produce an adequate sputum sample within 3 to 6 weeks prior to the start of study medication
* Be a current or ex-smoker who has a smoking history of at least 10 pack years at screening
* Meet tuberculosis(TB) screening criteria as: no history of latent or active TB, no signs or symptoms suggestive of active TB, have not had recent (within 3 months) close contact with a person with active TB, and no evidence of current, active TB or old, inactive TB

Exclusion criteria:

* Pulmonary disease, such as asthma, clinically significant bronchiectasis, cystic fibrosis, sarcoidosis, interstitial lung disorder, moderate or severe sleep apnea, or pulmonary hypertension at screening
* Has ever experienced life-threatening COPD, had a lung lobectomy, lung cancer surgery, lung volume reduction, or a lung transplant
* Requires oxygen therapy on a daily basis (greater than 12 hours/day) for chronic hypoxemia (inadequate level of oxygen in the blood) at screening
* Has received any live, attenuated viral or bacterial vaccines within 3 months prior to screening or is expected to receive any live attenuated vaccinations during the study or up to 6 months after the last administration of study medication
* Positive serology to human immunodeficiency virus 1 or 2, hepatitis B virus, or hepatitis C virus

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in prebronchodilator (before taking an inhaled bronchodilator) Forced Expiratory Volume in 1 second (FEV1) at Week 16 | Baseline (Week 0), Week 16
  FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.

SECONDARY OUTCOMES:
Change from baseline in postbronchodilator (after taking an inhaled bronchodilator) Forced Expiratory Volume in 1 second (FEV1) at Week 16 | Baseline (Week 0), Week 16
  FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.
Change from baseline in weekly average number of occasions in a day that rescue medication is used at Week 16 | Baseline (Week 0), Week 16
  Rescue medication is a relief medication for chronic obstructive pulmonary disease symptoms. e.g. when patients feel breathless, chest tight, or frequent cough. The reduction of number of the occasions indicates disease improvement with less symptoms.
Change from baseline in EXAcerbations of Chronic Pulmonary Disease Tool-Respiratory Symptoms™ (E-RS™) at Week 16 | Baseline (Week 0), Week 16
  E-RS is a 11-item respiratory system scoring algorithm to assess the severity of respiratory symptoms in participants with chronic obstructive pulmonary disease (COPD). Each item has either 5 or 6 response options. Higher score indicates more severe COPD.
Change from baseline at Week 16 in total score of the St George's respiratory questionnaire for Chronic Obstructive Pulmonary Disease (COPD) participants (SGRQ-C) | Baseline (Week 0), Week 16
  SGRQ-C is a 40-item questionnaire designed to measure health impairment in participants with COPD. SGRQ-C is divided into two components: 1) symptoms, 2) activity& impacts. Total SGRQ-C score ranges from 0 (best) and 100 (worst). Higher scores indicate greater health impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (44):
- Czechia (7):
  - Brno
  - Jindřichův Hradec
  - Karlovy Vary
  - Mělník
  - Prague
  - Praha 5 - Radotin
  - Strakonice
- Germany (8):
  - Berlin
  - Dresden
  - Frankfurt
  - Großhansdorf
  - Hanover
  - Koblenz
  - Magdeburg
  - Rüdersdorf
- Hungary (8):
  - Balassagyarmat
  - Budapest
  - Farkasgyepü
  - Komárom
  - Létavértes
  - Mohács
  - Nagykanizsa
  - Zalaegerszeg-P Zva N/A
- Malaysia (3):
  - Batu Caves
  - Kota Bharu
  - Kuala Lumpur
- Poland (4):
  - Krakow
  - Lodz
  - Poznan
  - Wroclaw
- Russia (9):
  - Barnaul
  - Kemerovo
  - Novosibirsk
  - Saint Petersberg
  - Saint Petersburg
  - Saint-Petersberg
  - Saratov
  - Yaroslavl
  - Yekaterinburg
- South Korea (3):
  - Seoul
  - Suwon
  - Wŏnju
- Taiwan (2):
  - New Taipei City
  - Taipei

REFERENCES:
- [Derived] Eich A, Urban V, Jutel M, Vlcek J, Shim JJ, Trofimov VI, Liam CK, Kuo PH, Hou Y, Xiao J, Branigan P, O'Brien CD. A Randomized, Placebo-Controlled Phase 2 Trial of CNTO 6785 in Chronic Obstructive Pulmonary Disease. COPD. 2017 Oct;14(5):476-483. doi: 10.1080/15412555.2017.1335697. Epub 2017 Jul 28. PMID 28753067